CLINICAL TRIAL: NCT06497088
Title: A Clinical Study to Evaluate the Ultrasonic Detection of a Novel Nasogastric Tube in the Human Body
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nasotrak Medical Pte Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NST-DHF-076
Record Dates: First submitted 2024-07-04; First posted 2024-07-11 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Nasogastric Tube Placement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Nasotrak System (Experimental)
  Interventions: Device: Nasotrak System

INTERVENTIONS:
Device: Nasotrak System — Device: The Nasotrak System
  The Nasotrak Medical System is intended to aid, in conjunction with institutional protocols, qualified operators in the placement of the Nasotrak's 12 Fr feeding tube into the stomach of patients requiring enteral feeding after insertion and before every feed. The Nasotrak nasogastric tube(NGT) is designed for use with Nasotrak's handheld device (HHD) which is able to detect the tip of the NGT via piezoelectric sensor, which converts ultrasound waves to electronic signals, thus assisting to track its location as an indicator of placement in the stomach. Nasotrak's NGT is intended only to be used with Nasotrak's HHD.
  The Nasotrak NGT is intended for the administration of nutrition, fluids and medications by the nasoenteric route for patients who have an intact gastrointestinal tract but are physically unable to manage nutritional intake through normal mastication and deglutition.

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy and accuracy of the Nasotrak System in an adult patient population.

ELIGIBILITY:
Inclusion Criteria:

* Adults greater than 18 years of age
* Able to provide informed consent or have a legally authorized representative available to provide informed consent in English
* Clinically requiring a 12 Fr NG/OG tube with X-ray confirmation per standard protocol

Exclusion Criteria:

* Female subjects of childbearing age with known pregnancy or lactating.
* Prisoners.
* Unable to consent in English.
* Subjects/ volunteers with pacemakers or life-sustaining devices in the body such as ICD.
* Subjects with a history of:
* Esophageal varices or ulcers.
* Upper airway obstruction.
* Upper GI stenosis or obstruction.
* Trauma involving sinuses, nares face or neck that would prevent nasogastric (NG) or oral tube insertion.
* Deformities of the sinus cavities and/or skull base.
* Esophageal cancer or neoplasm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effectiveness of detecting Nasotrak's nasogastric tube's distal tip using Nasotrak's ultrasound verification algorithm compared to X-ray. | 1 year
  All patients will receive placement verification per institutional practice

CONTACTS AND LOCATIONS:
Overall Officials: David Tan, Beng, Study Chair — Nasotrak Medical Pte Ltd
Locations (2):
- United States (2):
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Columbia University Medical Center, New York, New York